CLINICAL TRIAL: NCT04253613
Title: Laser Biostimulation in Periodontal Treatment of Diabetic and Systemically Healthy Periodontitis Patients
Brief Title: Laser Biostimulation in Periodontal Treatment
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, muge lutfioglu, Associate Professor, Ondokuz Mayıs University
Other Study IDs: OMU KAEK2012/49
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Inflammation; Periodontal Diseases
Keywords: periodontitis; diabetes mellitus; periodontal treatment; laser biostimulation therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- periodontal therapy: Systemically healthy subjects with periodontitis that have the sides treated with non-surgical periodontal treatment (NSPT) split-mouth designed study
- periodontal+laser therapy: Systemically healthy subjects with periodontitis that have the contra-lateral sides treated with laser biostimulation therapy(LBT) adjunct to non-surgical periodontal treatment(NSPT) split-mouth designed study
- diabetic periodontal therapy: Type 2 diabetic(DM2) subjects with periodontitis that have the sides treated with non-surgical periodontal treatment (NSPT) split-mouth designed study
- diabetic periodontal+laser therapy: Type 2 diabetic(DM2) subjects with periodontitis that have the contra-lateral sides treated with laser biostimulation therapy(LBT) adjunct to non-surgical periodontal treatment (NSPT) split-mouth designed study

SUMMARY:
The use of nonsurgical periodontal treatment, together with plaque control is considered the gold standart for the treatment of periodontal diseases; it produces beneficial effects such as reductions in clinical inflammation, decreases in pocket depth and increases in clinical attachment levels .However to modulate the healing response additional protocols has been suggested to increase the efficacy of existing treatment protocols. Laser biostimulation therapy is highly preferred method used due to its healing acceleration effect on several wounds in medical field. Thus,the investigators aimed to evaluate the laser biostimulation therapy adjunct to non-surgical periodontal treatment in systemically healthy and uncontrolled type 2 diabetes mellitus patients with generalized periodontitis. The effects of laser irradiation with Nd-YAG laser at the 1064-nm wavelength as an adjunct to non-surgical periodontal treatment (NSPT) was analysed by means of IL-1β and IL-10 concentrations in gingival crevicular fluid and periodontal clinical measurements of systemically healthy and uncontroled DM2 patients with generalized periodontitis.

DETAILED DESCRIPTION:
Today, the one that stands out the most among these protocols is laser application which was concluded to be a support or be an alternative treatment approach to standart periodontal treatments . As the laser biostimulation therapy(LBT) has been investigated by means of anti-inflammatory and healing promotion action on periodontal tissues, the LBT adjunct to non-surgical periodontal treatment of diabetic patients expected to create positive healing effects. The biostimulation effect of laser on tissue healing has drawn significant attention, not only in healthy individuals but also in patients with systemic problems causing impaired wound healing such as diabetes mellitus . Patients with poor metabolic control frequently present impaired wound healing and using LBT as a treatment method for diabetic ulcers have shown positive healing effects . However, there has been little knowledge about the additional benefits of LBT on healing proccess or inflammatory response among patients with uncontrolled diabetes mellitus type 2 receiving periodontal treatment.

In the light of the current knowledge, the impaired wound healing seen in diabetic patients may be a reason to require an additional approach in periodontal treatment like biostimulation of periodontal tissues by several ways. In order to determine the healing response, the investigators aimed to evaluate the effects of LBT irradiation with Nd-YAG laser at the 1064-nm wavelength as an adjunct to non-surgical periodontal treatment (NSPT) by means of periodontal clinical measurements and gingival crevicular fluid cytokine levels (IL-1β and IL-10) in systemically healthy and uncontroled DM2 patients with generalized periodontitis .

The study was designed as a split-mouth randomized, controlled, double-blind clinical study. The study protocol was approved by the Local Ethics Committee of Ondokuz Mayıs University and Turkey Ministry of Health, Drug and Medical Device Agency . The written informed consent was obtained from all study participants in accordance with the Helsinki Declaration .

All participants with periodontitis received NSPT. Non-surgical periodontal treatment consisted of conventional quadrant scaling in four session of 30 min, each on a weekly basis, using scalers, curettes and ultrasonic devices.

Laser Biostimulation treatment (LBT) and Sham application: Following NSPT, either the left or right side of each periodontitis patient was randomly selected (by coin toss) to receive LBT or sham treatment. LBT was performed six times (on the same day 30 which was the last scalling and root planning session and repeated weekly for 5 more times) using a 1064 nm Nd.YAG laser (Fotona AT Fidelis III,Ljubljana, Slovenia).

Clinical Measurements and Gingival creviculat fluid (GCF) Sampling Clinical measurements were performed before NSPT (baseline) and on days 30, 37 and 72 of the follow-up for both DM2 and SH groups. The following clinical periodontal measurements were recorded Silness & Löe plaque index (PI), Löe & Silness gingival index(GI), probing pocket depth (PPD); clinical attachment level (CAL); bleeding on probing (BOP). A Williams periodontal probe (Nordent Manufacturing Inc., Elk Grove Village, IL, USA) calibrated in mm was used to measure 6 sites on each selected tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual locations). For each tooth, the side with the highest PPD and CAL values were identified, and the additional clinical measurements and GCF sampling were performed on this side in both LBT and sham application of the patients. (total: 30 teeth in DM2 group, 30 teeth in SH group). GCF samples were collected before NSPT treatment(baseline) and on Days 30, 37 and 72 of follow-up. Sampling sites were isolated with cotton rolls, saliva was removed, and supragingival plaque, if present, was removed using a sterile curette. GCF was sampled by placing a strip of filter paper (Periopaper, ProFlow, Inc., Amityville, New York, USA) into the crevice until mild resistance was felt and then leaving it in position for 30 seconds. The GCF volume of each strip was determined by electronic impedance (Periotron 8000, ProFlow, Inc.), and samples were then placed in sterile polypropylene tubes and stored at -70°C until analysis.

Amounts of IL-1β and IL-10 in each GCF sample were evaluated using standard enzyme-linked immunosorbent assays (ELISA) according to the manufacturers' instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study, being male and ≥ 35 years of age,
2. Having been diagnosed as type 2 diabates mellitus (DM2) with the ADA criteria at least 2 years before the study and having an HbA1c value of ≥ 7 for DM2 group,
3. Not having a systemic disease other than DM2 for diabetic group; and not having any systemical diseases for systemically healthy group,
4. Not having any systemic complications of diabetes,
5. Not smoking or consuming alcohol,
6. Having at least 20 teeth,
7. Having at least two single-rooted teeth (like one premolar or incisor tooth) representing symmetrical or same group teeth with gingival index≥2, bleeding on probing (+), probing pocket depth and/or clinical attachment lvel >5 mm as well as ≥30% radiographically observable alveolar bone loss, on the left and right area of mandibular,
8. Being able to fulfill the instructions for oral hygiene training

Exclusion Criteria:

1. using systemic antimicrobials, non-steroidal anti-inflammatory drugs and/or steroids during the 6 weeks prior to data collection
2. received periodontal treatment in the 6 months prior to data collection
3. having predisposing factors such as a dental crown, bridge, filling, or cavity on teeth from which the GCF was to be collected.

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was designed as a split-mouth, controlled, double-blind clinical study. Participants were recruited among patients admitted to the periodontology clinic in Ondokuz Mayıs university Dental Faculty. Periodontal status was assessed and diagnosed as generalized periodontitis. In the mouth of each patient in both diabetic and healthy population, two symmetrical teeth were assigned as one side to apply non-surgical periodontal treatment alone and the other side to apply laser biostimulation therapy adjunct to NSPT. Thus,15 diabetic and 15 systemically helathy subjects included in the split-mouth designed study and 4 groups were constituted as:periodontal therapy (n=15, Split-mouth); periodontal+laser therapy (n=15, Split-mouth); diabetic periodontal therapy (n=15, Split-mouth); diabetic periodontal+laser therapy(n=15, Split-mouth):
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2014-06-15 (Actual); Study Completion 2014-06-15 (Actual)

PRIMARY OUTCOMES:
IL-1β level in GCF | GCF sampling was performed prior to periodontal treatment and on days 30,37,72 of follow-up.
  IL-1β is a cytokine present in gingival crevicular fluid (GCF). Its concentration is calculated as picogram/microliter and it changes due to the elimination of inflammation by periodontal therapy.
IL-10 level in GCF | GCF sampling was performed prior to periodontal treatment and on days 30,37,72 of follow-up.
  IL-10 is a cytokine present in gingival crevicular fluid (GCF). Its concentration is calculated as picogram/microliter and it changes due to the elimination of inflammation by periodontal therapy.

IPD SHARING:
Plan to Share IPD: No